CLINICAL TRIAL: NCT04239638
Title: Analysis of Cervical Spinal MRI With Deep Learning
Status: Withdrawn | Type: Observational
Why Stopped: postponed to a later date
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 54022451
Record Dates: First submitted 2020-01-15; First posted 2020-01-27 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Cervical Disc Disease; Cervical Spine Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — MRI images
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cervical Spinal MRI — Cervical Spinal MRI images of 500 patients will be entered into the system for modeling

SUMMARY:
The aim of this study is analyzing the pathologies in cervical spinal MRI images by using image processing algorithms. Determination of these pathological cases which taught to the system with deep learning and determination of their levels. Finally; verification of the system by comparing radiologist reports and automated system outputs.

DETAILED DESCRIPTION:
Neck pain is a very common health problem with a worldwide prevalence ranging from 16.7% to 75.1%. The source of neck pain is often considered - although there is no strong evidence - the cervical intervertebral disc. Radiological imaging methods are used for the detection of degeneration of the discs and the end plaque changes in the vertebral body corresponding to this degeneration.Magnetic Resonance Imaging (MRI) gives information about the structure of intervertebral disc, width of spinal canal and tissues outside the canal. However, there is no standardization in the identification and evaluation of radiological images, and interobserver variability is high. Studies have been initiated on automated systems that analyze MRI images to increase the accuracy and consistency of reporting procedures. Examining MRI images with deep learning can lead to the production of systems that help clinical decision making and also allows the evaluation of large data in a short time.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Having result of a cervical spinal MRI, which was performed for neck pain in the hospital records in the last 5 years.

Exclusion Criteria:

* Malignancy
* Signs of active infection
* Significant spinal vertebral deformity (advanced scoliosis, congenital vertebral defects)
* Spinal surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with neck pain between 18-75 years
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy rate of the model as assessed by cross validation of the data set | Through study completion, an average of 1,5 years
  We will randomly divide the dataset into 4 subsets. In each sub-experiments, MRI slices from 3 subsets will be trained and slices in the other subset will be tested. We will perform totally 4 sub-experiments, so each slice in the dataset will be tested once.
Reliability of the model as assessed by comparing the reports of the model and radiologist. | Through study completion, an average of 1,5 years
  Kappa statistics and reliability coefficients will be use.

CONTACTS AND LOCATIONS:
Overall Officials: Bugra Ince, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Castro-Mateos I, Hua R, Pozo JM, Lazary A, Frangi AF. Intervertebral disc classification by its degree of degeneration from T2-weighted magnetic resonance images. Eur Spine J. 2016 Sep;25(9):2721-7. doi: 10.1007/s00586-016-4654-6. Epub 2016 Jul 7. PMID 27388019
- [Background] Jamaludin A, Lootus M, Kadir T, Zisserman A, Urban J, Battie MC, Fairbank J, McCall I; Genodisc Consortium. ISSLS PRIZE IN BIOENGINEERING SCIENCE 2017: Automation of reading of radiological features from magnetic resonance images (MRIs) of the lumbar spine without human intervention is comparable with an expert radiologist. Eur Spine J. 2017 May;26(5):1374-1383. doi: 10.1007/s00586-017-4956-3. Epub 2017 Feb 6. PMID 28168339
- [Background] Kim S, Bae WC, Masuda K, Chung CB, Hwang D. Fine-Grain Segmentation of the Intervertebral Discs from MR Spine Images Using Deep Convolutional Neural Networks: BSU-Net. Appl Sci (Basel). 2018 Sep;8(9):1656. doi: 10.3390/app8091656. Epub 2018 Sep 14. PMID 30637135
- [Background] Daenzer S, Freitag S, von Sachsen S, Steinke H, Groll M, Meixensberger J, Leimert M. VolHOG: a volumetric object recognition approach based on bivariate histograms of oriented gradients for vertebra detection in cervical spine MRI. Med Phys. 2014 Aug;41(8):082305. doi: 10.1118/1.4890587. PMID 25086554